CLINICAL TRIAL: NCT03771456
Title: Anastomotic Leakage and Enhanced Recovery Pathways After Colorectal Surgery: the Italian ColoRectal Anastomotic Leakage Study Group (iCral 2)
Brief Title: Anastomotic Leakage and Enhanced Recovery Pathways After Colorectal Surgery
Acronym: iCral2
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ospedale C & G Mazzoni (Other)
Responsible Party: Principal Investigator, Marco Catarci, Director, General Surgery Unit, Ospedale C & G Mazzoni
Other Study IDs: 2.0
Record Dates: First submitted 2018-12-06; First posted 2018-12-11 (Actual); Last update posted 2018-12-11 (Actual); Status verified 2018-12

CONDITIONS: Colorectal Neoplasms; Anastomotic Leak; Surgery--Complications
MeSH Terms: conditions — Colorectal Neoplasms; Anastomotic Leak

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Procedure: Colorectal resections — Colorectal resections

SUMMARY:
Prospective observational multicenter study on the influence of adherence to enhanced recovery pathways on early outcomes (anastomotic leakage, morbidity, mortality, readmission, reoperation rates and length of postoperative stay) after elective colorectal surgery in Italy.

DETAILED DESCRIPTION:
BACKGROUND

Anastomotic leakage (AL) is a dreaded major complication after colorectal surgery. The overall incidence of anastomotic dehiscence and subsequent leaks is 2 to 7 percent when performed by experienced surgeons. The lowest leak rates are found with ileocolic anastomoses (1 to 3 percent) and the highest occur with coloanal anastomosis (10 to 20 percent). Leaks usually become apparent between five and seven days postoperatively. Almost half of all leaks occur after the patient has been discharged, and up to 12 percent occur after postoperative day (POD) 30. Late leaks often present insidiously with low-grade fever, prolonged ileus, and nonspecific symptoms attributable to other postoperative infectious complications. Small, contained leaks present later in the clinical course and may be difficult to distinguish from postoperative abscesses by radiologic imaging, making the diagnosis uncertain and underreported.

There is no uniform definition of an anastomotic dehiscence and leak. In a review of 97 studies, as an example, 56 different definitions of an anastomotic leak were used. The majority of reports define an anastomotic leak using clinical signs, radiographic findings, and intraoperative findings. The clinical signs include: Pain, Fever, Tachycardia, Peritonitis, Feculent drainage, Purulent drainage. The radiographic signs include: Fluid collections, Gas containing collections. The intraoperative findings include: Gross enteric spillage, Anastomotic disruption.

Risk factors for a dehiscence and leak are classified according to the site of the anastomosis (extraperitoneal or intraperitoneal). A prospective review of 1598 patients undergoing 1639 anastomotic procedures for benign or malignant colorectal disease found a significantly increased risk of anastomotic leak with extraperitoneal compared with intraperitoneal anastomoses (6.6 versus 1.5 percent; 2.4 percent overall).

Major risk factors for an extraperitoneal AL include: The distance of the anastomosis from the anal verge (Patients with a low anterior resection and an anastomosis within 5 cm from the anal verge are the highest risk group for an anastomotic leak), Anastomotic ischemia, Male gender, Obesity.

Major risk factors for an intraperitoneal AL include: American Society of Anesthesiologists (ASA) score Grade III to V, Emergent surgery, Prolonged operative time, Hand-sewn ileocolic anastomosis.

Controversial, inconclusive, or pertinent negative associations between the following variables and AL have been reported: Neoadjuvant radiation therapy, Drains, Protective stoma, Hand-sewn colorectal anastomosis, Laparoscopic procedure, Mechanical bowel preparation, Nutritional status, Perioperative corticosteroids.

Enhanced Recovery After Surgery (ERAS) programs for colorectal surgery have been extensively studied during the last 20 years. It is now clear that they offer a consistent reduction of overall morbidity rates, postoperative length of stay and costs, and that there is a clear dose-effect relation between adherence to at least 60-70% of the program items and these outcomes. On the other hand, little is known concerning the potential benefit of ERAS programs over AL rates or if adherence to specific items of the program may reduce AL rates.

Therefore, the investigators planned this study to prospectively evaluate AL rates after colorectal resections and their interaction with known risk factors and ERAS program items.

METHODS

Prospective enrollment from January to December 2019 in 41 Italian surgical centers. All patients undergoing elective colorectal surgery with anastomosis will be included in a prospective database after having provided a written informed consent. A total of 1,750 patients is expected based on a mean of 43 cases/year per center.

Outcome measures

1. Preoperative risk factors of anastomotic leakage (age, gender, obesity, nutritional status, diabetes, cardiovascular disease, chronic liver disease, renal failure, inflammatory bowel disease, perioperative steroid therapy, ASA class I-II vs III)
2. Operative parameters (approach, procedure, anastomotic technique, length of operation, disease stage)
3. ERAS program items (prehabilitation, counseling, nutritional evaluation, immuno-nutrition, deep venous thrombosis prophylaxis, antibiotic prophylaxis, bowel preparation, preoperative carbohydrates load, standardized anesthesia protocol, restrictive i.v. fluid administration, control of body temperature, nausea and vomit prophylaxis, multimodal approach to opioid-sparing pain control, restrictive use of surgical drains, laparoscopic surgery, removal of nasogastric tubes before reversal of anesthesia, early removal of urinary catheter, early mobilization, early oral intake of fluids and solids, use of chewing gums and laxatives, intake of protein-rich nutritional supplements, prepare for early discharge, audit).

Endpoints

1. Anastomotic leakage rate
2. Minor and major complications
3. Length of postoperative hospital stay
4. Readmission and reoperation rates Recorded data and follow-up Potential patient-specific and intraoperative risk factors will be recorded: gender, body mass index, nutritional status according to the Mini Nutritional Assessment short-form, surgical indication (cancer, polyps, chronic inflammatory bowel disease, diverticular disease), preoperative albuminemia, use of steroids, renal failure and dialysis, cardiovascular or respiratory disease, American Society of Anesthesia class, bowel preparation (decision made by operating surgeon), laparoscopy or laparotomy, level of anastomosis and technique (mechanical or hand-sewn, intra- or extra-corporeal), operative time, presence of drainage, and perioperative blood transfusion(s). During the postoperative period, patients will be examined by the attending surgeon daily. Fever (central temperature > 38 °C), pulse, abdominal signs, bowel movements, volume and aspect of drainage (if present) will be recorded daily. The attending surgeon will make any decision for complementary exams and imaging according to his own criteria. The rate of any complication will be calculated and graded including all leaks (independently of clinical significance), wound infection (according to the definitions of the Centers for Disease Control and Prevention and wound culture), pneumonia (clinical symptoms, and physical and radiological examinations), central line infection (positive blood culture), urinary tract infection (positive urine culture with bacterial count ). Patients will be followed-up in the outpatient clinic up to 6 weeks after discharge from the hospital.

Main endpoint is anastomotic dehiscence (intended as any deviation from the planned postoperative course related to the anastomosis, or presence of pus or enteric contents within the drains, presence of abdominal or pelvic collection in the area of the anastomosis on postoperative CT scan, performed at the discretion of the attending surgeon, leakage of contrast through the anastomosis during enema or evident anastomotic dehiscence at reoperation for postoperative peritonitis). Thus, all detected leaks will be considered independently of clinical significance. No imaging will be performed routinely in order to search for leakage.

Secondary endpoints are morbidity and mortality rates, postoperative length of stay, readmission and reoperation rates.

After anonymization, all data of each single case will be prospectively uploaded by every local investigator on a protected web-based database. Thereafter, all data will be incorporated into a spreadsheet (MS Excel) for data analysis, checking for any discrepancy, that will be addressed and solved through strict cooperation between chief investigator, data manager and participating center.

Statistical Analysis Quantitative values will be expressed as mean ± standard deviation, median and range; categorical data with percentage frequencies. Mean values of duration of stay will be compared according to the presence or absence of fistulas using Student's two-sided t test (allowing for heterogeneity of variances) or with a non-parametric Mann-Whitney test. Both univariate analysis and multivariate analysis will be performed to assess risk factors for leakage and overall complications. The odds ratio (OR) will be presented followed by its 95% confidence interval (95% CI). For all statistical tests the significant level is fixed at p < .05.

Statistical analyses will be carried out using STATA software (Stata Corp. College Station, Texas, USA).

Sample size Considering that adherence to 70% of the items of an ERAS program determines a significant reduction in surgical complications after colorectal surgery, an estimation of the OR for AL and ERAS program adherence at 70% of the items is equal to 0.55 (95% c.i. 0.36-0.87); assuming a maximum error equal to 0.04, the required sample size is n=1,748 (about 874 cases per arm expected in low vs high adherence to ERAS programs).

ELIGIBILITY:
Inclusion Criteria:

1. Patients submitted to laparoscopic/robotic/open/converted ileo-colo-rectal resection with anastomosis (both intra- and extra-corporeal), including planned Hartmann's reversals.
2. American Society of Anesthesiologists' (ASA) class I, II or III
3. Elective or delayed urgency surgery
4. Patients' written acceptance to be included in the study.

Exclusion Criteria:

1. American Society of Anesthesiologists' (ASA) class IV-V
2. Patients with stoma before or at operation
3. Simple stoma closure
4. Transanal procedure
5. Pregnancy
6. Hyperthermic intraperitoneal chemotherapy for carcinomatosis.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any patient submitted to elective colorectal resection with anastomosis
Sampling Method: Non-Probability Sample
Enrollment: 1748 (Estimated)
Dates: Start 2019-01-07 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Anastomotic Leakage rate | up to 45 days
  Rate of any complication related to the anastomosis after colorectal resection

SECONDARY OUTCOMES:
Morbidity rate | up to 45 days
  Rate of any complication after colorectal resection
Mortality rate | up to 45 days
  Rate of any death after colorectal resection
Reoperation rate | up to 45 days
  Rate of any unplanned reoperation
Readmission rate | up to 45 days
  Rate of any unplanned readmission after discharge
Length of postoperative hospital stay | up to 45 days
  number of days between primary colorectal resection and discharge

CONTACTS AND LOCATIONS:
Overall Officials: Marco Catarci, MD FACS, Study Chair — Ospedale C & G Mazzoni - Ascoli Piceno; Gianluca Guercioni, MD, Principal Investigator — Ospedale C & G Mazzoni - Ascoli Piceno
Locations (41):
- Italy (41):
  - UOC Chirurgia Generale - Ospedale Profili - Fabriano (AN) - ASUR MARCHE AV2, Fabriano, AN
  - UOC Chirurgia Generale - Ospedale "C. Urbani" Jesi - AV2 - ASUR Marche, Iesi, AN
  - UOC Chirurgia Generale e d'Urgenza - Ospedale Regionale "U. Parini" - Aosta, Aosta, AO
  - UOC Chirurgia Generale - Ascoli Piceno - AV5 - ASUR Marche, Ascoli Piceno, AP
  - UOC Chirurgia Generale - San Benedetto del Tronto (AP) - AV5 - ASUR Marche, San Benedetto del Tronto, AP
  - UOC Chirurgia Generale Universitaria - Ospedale San Salvatore - L'Aquila, L’Aquila, AQ
  - UOC Chirurgia Oncologica - AORN San Giuseppe Moscati - Avellino, Avellino, AV
  - Clinica Chirurgica, Università di Brescia - UOC Chirurgia Generale 3, ASST Spedali Civili di Brescia - Brescia, Brescia, BS
  - UOC Chirurgia Generale - Ospedale Montichiari (BS) - ASST Spedali Civili di Brescia, Montichiari, BS
  - S.C. Chirurgia Generale e Oncologica - Azienda Ospedaliera S. Croce e Carle - Cuneo, Italia, Cuneo, CN
  - UOC Chirurgia Generale 1 - Chirurgia laparoscopica - Università di Ferrara, Ferrara, FE
  - UOC di Chirurgia Addominale IRCCS Casa Sollievo della Sofferenza - San Giovanni Rotondo - Foggia, San Giovanni Rotondo, FG
  - UOC Chirurgia Generale - Ospedale S. Maria Annunziata - Firenze - ASL Toscana Centro, Florence, FI
  - UOC Chirurgia Generale ad Indirizzo Oncologico - IRCCS San Martino IST - Genova, Genova, GE
  - UOC Chirurgia Generale - Ospedale"San Giovanni di Dio", ASP di Crotone (KR), Crotone, KR
  - UOC Chirurgia Generale e d'Urgenza - Ospedale Cardinale Panico - Tricase (LE), Tricase, LE
  - UOC Chirurgia Generale - ASST Nord - Sesto San Giovanni (MI), Sesto San Giovanni, MI
  - UOC Chirurgia Generale - Ospedale di Esine (BS) - ASST Valcamonica, Esine, NS
  - UOC Chirurgia Generale e D'Urgenza - Pescara, Pescara, PE
  - UOC Chirurgia Generale - Foligno (PG) - USL UMBRIA 2, Foligno, PG
  - SC Chirurgia Generale e Oncologica - AO Marche Nord - Pesaro, Pesaro, PU
  - UOC Chirurgia Generale - Ragusa, Ragusa, RG
  - UOC Chirurgia Generale - Ospedale "Regina Apostolorum" Albano Laziale (RM), Albano Laziale, RM
  - UOC Chirurgia Generale e d'Urgenza - Policlinico Casilino - Roma, Roma, RM
  - UOC Chirurgia Generale e D'Urgenza . Azienda Ospedaliera San Camillo Forlanini Roma, Roma, RM
  - UOC Chirurgia Generale e Oncologica - Ospedale San Filippo Neri - ASL Roma1, Roma, RM
  - UOS Chirurgia Geriatrica - Università Campus BioMedico - Roma, Roma, RM
  - UOSD Chirurgia Mininvasiva e dell'Apparato Digerente - Università Tor Vergata - Roma, Roma, RM
  - UOC Chirurgia Generale, Ospedale "Ceccarini" di Riccione (RN), Riccione, RN
  - UOC Chirurgia Generale e d'urgenza, Rimini, Novafeltria, Santarcangelo, Rimini, RN
  - UOC Chirurgia Generale I - Ospedale di La Spezia - ASL5 Spezzino, La Spezia, SP
  - UOC Chirurgia Generale 1 - Ospedale S. Chiara - APSS Trento, Trento, TN
  - UOC Chirurgia Generale e Mininvasiva, Ospedale San Camillo di Trento, Trento, TN
  - UOC Chirurgia Generale - Ospedale "E. Agnelli" di Pinerolo (TO) - ASL TO3, Pinerolo, TO
  - UOC Chirurgia Generale - Conegliano Veneto (TV) AULSS2 Marca trevigiana, Conegliano, TV
  - UOC Chirurgia Generale - Ospedale Sacro Cuore Don Calabria Negrar Verona, Negrar, VR
  - U.O.C. di Chirurgia Generale e dell'Esofago e Stomaco - AOUI di Verona, Verona, VR
  - UOC Chirurgia Generale Epatobiliare - AOUI Verona, Verona, VR
  - UOC Chirurgia Generale Oncologica - Azienda Ospedaliera Belcolle - Viterbo, Viterbo, VT
  - SOC Chirurgia Colorettale - Istituto Nazionale dei Tumori - IRCCS Fondazione "G.Pascale" - Napoli, Napoli
  - UOC Chirurgia Generale - Pozzuoli (NA) - ASL Napoli2 nord, Pozzuoli

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Boushey R, Williams LJ. Management of anastomotic complications of colorectal surgery. Uptodate 2017.
- [Background] Slieker JC, Komen N, Mannaerts GH, Karsten TM, Willemsen P, Murawska M, Jeekel J, Lange JF. Long-term and perioperative corticosteroids in anastomotic leakage: a prospective study of 259 left-sided colorectal anastomoses. Arch Surg. 2012 May;147(5):447-52. doi: 10.1001/archsurg.2011.1690. PMID 22249852
- [Background] Kingham TP, Pachter HL. Colonic anastomotic leak: risk factors, diagnosis, and treatment. J Am Coll Surg. 2009 Feb;208(2):269-78. doi: 10.1016/j.jamcollsurg.2008.10.015. Epub 2008 Dec 4. No abstract available. PMID 19228539
- [Background] Hyman N, Manchester TL, Osler T, Burns B, Cataldo PA. Anastomotic leaks after intestinal anastomosis: it's later than you think. Ann Surg. 2007 Feb;245(2):254-8. doi: 10.1097/01.sla.0000225083.27182.85. PMID 17245179
- [Background] Park JS, Choi GS, Kim SH, Kim HR, Kim NK, Lee KY, Kang SB, Kim JY, Lee KY, Kim BC, Bae BN, Son GM, Lee SI, Kang H. Multicenter analysis of risk factors for anastomotic leakage after laparoscopic rectal cancer excision: the Korean laparoscopic colorectal surgery study group. Ann Surg. 2013 Apr;257(4):665-71. doi: 10.1097/SLA.0b013e31827b8ed9. PMID 23333881
- [Background] Dietz, DW, Bailey, HR. Postoperative complications. In: ASCRS Textbook of Colon and Rectal Surgery, Church, JM, Beck, DE, Wolff, BG, Fleshman, JW, Pemberton, JH, (Eds), Springer-Verlag New York, LLC, New York 2006. p.141.
- [Background] Bruce J, Krukowski ZH, Al-Khairy G, Russell EM, Park KG. Systematic review of the definition and measurement of anastomotic leak after gastrointestinal surgery. Br J Surg. 2001 Sep;88(9):1157-68. doi: 10.1046/j.0007-1323.2001.01829.x. PMID 11531861
- [Background] Law WI, Chu KW, Ho JW, Chan CW. Risk factors for anastomotic leakage after low anterior resection with total mesorectal excision. Am J Surg. 2000 Feb;179(2):92-6. doi: 10.1016/s0002-9610(00)00252-x. PMID 10773140
- [Background] Lipska MA, Bissett IP, Parry BR, Merrie AE. Anastomotic leakage after lower gastrointestinal anastomosis: men are at a higher risk. ANZ J Surg. 2006 Jul;76(7):579-85. doi: 10.1111/j.1445-2197.2006.03780.x. PMID 16813622
- [Background] Platell C, Barwood N, Dorfmann G, Makin G. The incidence of anastomotic leaks in patients undergoing colorectal surgery. Colorectal Dis. 2007 Jan;9(1):71-9. doi: 10.1111/j.1463-1318.2006.01002.x. PMID 17181849
- [Background] Ljungqvist O, Scott M, Fearon KC. Enhanced Recovery After Surgery: A Review. JAMA Surg. 2017 Mar 1;152(3):292-298. doi: 10.1001/jamasurg.2016.4952. PMID 28097305
- [Background] Ljungqvist O, Thanh NX, Nelson G. ERAS-Value based surgery. J Surg Oncol. 2017 Oct;116(5):608-612. doi: 10.1002/jso.24820. Epub 2017 Sep 5. PMID 28873501
- [Background] Nelson G, Kiyang LN, Crumley ET, Chuck A, Nguyen T, Faris P, Wasylak T, Basualdo-Hammond C, McKay S, Ljungqvist O, Gramlich LM. Implementation of Enhanced Recovery After Surgery (ERAS) Across a Provincial Healthcare System: The ERAS Alberta Colorectal Surgery Experience. World J Surg. 2016 May;40(5):1092-103. doi: 10.1007/s00268-016-3472-7. PMID 26928854
- [Background] Neville A, Lee L, Antonescu I, Mayo NE, Vassiliou MC, Fried GM, Feldman LS. Systematic review of outcomes used to evaluate enhanced recovery after surgery. Br J Surg. 2014 Feb;101(3):159-70. doi: 10.1002/bjs.9324. PMID 24469616
- [Background] ERAS Compliance Group. The Impact of Enhanced Recovery Protocol Compliance on Elective Colorectal Cancer Resection: Results From an International Registry. Ann Surg. 2015 Jun;261(6):1153-9. doi: 10.1097/SLA.0000000000001029. PMID 25671587
- [Background] Gustafsson UO, Scott MJ, Schwenk W, Demartines N, Roulin D, Francis N, McNaught CE, Macfie J, Liberman AS, Soop M, Hill A, Kennedy RH, Lobo DN, Fearon K, Ljungqvist O; Enhanced Recovery After Surgery (ERAS) Society, for Perioperative Care; European Society for Clinical Nutrition and Metabolism (ESPEN); International Association for Surgical Metabolism and Nutrition (IASMEN). Guidelines for perioperative care in elective colonic surgery: Enhanced Recovery After Surgery (ERAS((R))) Society recommendations. World J Surg. 2013 Feb;37(2):259-84. doi: 10.1007/s00268-012-1772-0. No abstract available. PMID 23052794
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Background] Clavien PA, Barkun J, de Oliveira ML, Vauthey JN, Dindo D, Schulick RD, de Santibanes E, Pekolj J, Slankamenac K, Bassi C, Graf R, Vonlanthen R, Padbury R, Cameron JL, Makuuchi M. The Clavien-Dindo classification of surgical complications: five-year experience. Ann Surg. 2009 Aug;250(2):187-96. doi: 10.1097/SLA.0b013e3181b13ca2. PMID 19638912
- [Background] Kaiser MJ, Bauer JM, Ramsch C, Uter W, Guigoz Y, Cederholm T, Thomas DR, Anthony P, Charlton KE, Maggio M, Tsai AC, Grathwohl D, Vellas B, Sieber CC; MNA-International Group. Validation of the Mini Nutritional Assessment short-form (MNA-SF): a practical tool for identification of nutritional status. J Nutr Health Aging. 2009 Nov;13(9):782-8. doi: 10.1007/s12603-009-0214-7. PMID 19812868
- [Background] Skipper A, Ferguson M, Thompson K, Castellanos VH, Porcari J. Nutrition screening tools: an analysis of the evidence. JPEN J Parenter Enteral Nutr. 2012 May;36(3):292-8. doi: 10.1177/0148607111414023. Epub 2011 Nov 1. PMID 22045723
- [Background] Horan TC, Gaynes RP, Martone WJ, Jarvis WR, Emori TG. CDC definitions of nosocomial surgical site infections, 1992: a modification of CDC definitions of surgical wound infections. Infect Control Hosp Epidemiol. 1992 Oct;13(10):606-8. No abstract available. PMID 1334988
- [Derived] Catarci M, Ruffo G, Viola MG, Garulli G, Pavanello M, Scatizzi M, Bottino V, Guadagni S; Italian ColoRectal Anastomotic Leakage (iCral) study group. Enhanced Recovery Independently Lowers Failure to Rescue After Colorectal Surgery. Dis Colon Rectum. 2025 May 1;68(5):616-626. doi: 10.1097/DCR.0000000000003655. Epub 2025 Feb 11. PMID 39932201